CLINICAL TRIAL: NCT00138229
Title: Phase II Trial Using Aldesleukin (IL-2) Following a Lymphodepleting Chemotherapy and Reinfusion of Autologous Lymphocytes Depleted of T Regulatory Lymphocytes in Metastatic Melanoma
Brief Title: Cyclophosphamide and Fludarabine Followed By an Autologous Lymphocyte Infusion and Interleukin-2 in Treating Patients With Refractory or Recurrent Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 050194; 05-C-0194; NCI-P6573; CDR0000440165; NCT00118599 (obsolete NCT alias)
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Filgrastim; Cyclophosphamide; fludarabine phosphate

INTERVENTIONS:
Biological: aldesleukin
Biological: filgrastim
Biological: therapeutic autologous lymphocytes
Drug: cyclophosphamide
Drug: fludarabine phosphate

SUMMARY:
RATIONALE: An infusion of a patient's lymphocytes that have been treated in the laboratory to remove certain immune cells may be an effective treatment for melanoma. Drugs, such as cyclophosphamide and fludarabine, may suppress the immune system so that the patient's immune cells allow the infused lymphocytes to work. Interleukin-2 may help the lymphocytes kill more tumor cells when they are put back in the body. Giving cyclophosphamide and fludarabine followed by an autologous lymphocyte infusion and interleukin-2 may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cyclophosphamide and fludarabine followed by an autologous lymphocyte infusion and interleukin-2 works in treating patients with refractory or recurrent melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine tumor regression in patients with metastatic melanoma treated with nonmyeloablative lymphodepleting chemotherapy comprising cyclophosphamide and fludarabine followed by autologous CD25-positive-T-regulatory-cell-depleted lymphocyte reinfusion and high-dose interleukin-2.

Secondary

* Determine the rate of repopulation of CD25-positive T-regulatory cells in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE:

* Apheresis and CD25-positive T-regulatory cell depletion: Patients undergo 1-2 aphereses to collect peripheral blood mononuclear cells (PBMC). CD25-positive T-regulatory cells are depleted from the collected PBMC in vitro.
* Nonmyeloablative lymphodepleting chemotherapy: Patients receive cyclophosphamide IV over 1 hour on days -8 and -7 and fludarabine IV over 15-30 minutes on days -6 to -2.
* Autologous CD25-positive-T-regulatory-cell-depleted lymphocyte reinfusion: Patients receive autologous lymphocytes IV over 20-30 minutes on day 0.
* Filgrastim (G-CSF) and high-dose interleukin-2 (IL-2) therapy: Patients receive G-CSF subcutaneously (SC) daily beginning on day 0 and continuing until blood counts recover. Patients also receive high-dose IL-2 IV over 15 minutes 3 times daily on days 0-4 and 14-18. Patients are reevaluated 4-6 weeks after completion of high-dose IL-2 therapy. Patients achieving stable disease or a partial response may receive additional high-dose IL-2 as above for up to 2 retreatment courses in the absence of disease progression or unacceptable toxicity. Retreatment begins at least 6 weeks after autologous lymphocyte reinfusion.

After completion of study treatment, patients are followed at 4-6 weeks and then every 1-2 months thereafter.

PROJECTED ACCRUAL: A total of 16-29 patients will be accrued for this study within 1-1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of melanoma

  * Metastatic disease
* Measurable disease
* HLA-A2 negative disease
* Disease did not respond to OR recurred after completion of prior high-dose interleukin-2 (IL-2)
* Eligible to receive high-dose IL-2
* No tumor reactive cells available for cell transfer therapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 8.0 g/dL
* No coagulation disorders

Hepatic

* ALT and AST < 3 times upper limit of normal
* Bilirubin ≤ 2.0 mg/dL (< 3.0 mg/dL if due to Gilbert's syndrome)
* Hepatitis B surface antigen negative
* Hepatitis C antigen negative

Renal

* Creatinine ≤ 2.0 mg/dL
* No renal failure requiring dialysis due to toxic effects of prior IL-2 administration

Cardiovascular

* No myocardial infarction
* No cardiac arrhythmias
* No other major cardiovascular illness as evidenced by a positive stress thallium or comparable test
* Normal cardiac stress test (e.g., stress thallium, stress MUGA, dobutamine echocardiogram) AND LVEF ≥ 45% (for patients ≥ 50 years of age or who have a history of EKG abnormalities, symptoms of cardiac ischemia, or arrhythmias)

Pulmonary

* No obstructive or restrictive pulmonary disease
* No other major respiratory illness
* FEV_1 ≥ 60% of predicted (for patients with a prolonged history of cigarette smoking or symptoms of respiratory dysfunction)

Immunologic

* HIV negative
* Epstein-Barr virus positive
* No active systemic infection
* No autoimmune disease (e.g., autoimmune colitis or Crohn's disease)
* No immunodeficiency due to prior chemotherapy or radiotherapy

  * Recovered immune competence after prior chemotherapy or radiotherapy as evidenced by normal lymphocyte count and WBC and an absence of opportunistic infection
* No other major immune system disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 months after completion of study treatment
* No other toxic effects during prior IL-2 administration that would preclude redosing with IL-2, including the following:

  * Mental status changes that would require intubation
  * Bowel perforation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* At least 4 weeks since prior systemic therapy

Chemotherapy

* At least 6 weeks since prior nitrosoureas
* At least 4 weeks since prior systemic therapy

Endocrine therapy

* No concurrent systemic steroid therapy

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-07; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Tumor regression

SECONDARY OUTCOMES:
Rate of repopulation of CD25-positive T-regulatory cells
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Principal Investigator — NCI - Surgery Branch
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - NCI - Surgery Branch, Bethesda, Maryland